CLINICAL TRIAL: NCT00203892
Title: A Randomized Pilot Phase II Study of Immunization With Modified CEA (CAP1-6D) Peptide In Patients With Locally Advanced Or Surgically Resected Adenocarcinoma of the Pancreas
Brief Title: Study of CAP1-6D in Patients With Locally Advanced or Surgically Resected Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12095B
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Adenocarcinoma; Pancreas
MeSH Terms: conditions — Adenocarcinoma | interventions — CAP1-6D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: CEA peptide 10mcg (Experimental): Vaccine contained the modified CEA peptide (10mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Interventions: Biological: modified CEA peptide (10mcg)
- B: CEA peptide 100 mcg (Experimental): Vaccine contained the modified CEA peptide (100mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Interventions: Biological: modified CEA peptide (100mcg)
- C: CEA peptide 1000mcg (Experimental): Vaccine contained the modified CEA peptide (1000mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Interventions: Biological: modified CEA peptide (1000mcg)

INTERVENTIONS:
Biological: modified CEA peptide (10mcg) — Vaccine contained the modified CEA peptide (10mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Other Names: CAP1-6D
  Arms: A: CEA peptide 10mcg
Biological: modified CEA peptide (100mcg) — Vaccine contained the modified CEA peptide (100mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Other Names: CAP1-6D
  Arms: B: CEA peptide 100 mcg
Biological: modified CEA peptide (1000mcg) — Vaccine contained the modified CEA peptide (1000mcg), Montanide ISA-51, and sargramostim (GM-CSF) 250mcg. Vaccine was administered on Day 1 of each 14 day cycle until progressive disease or dose-limiting toxicity for a maximum of 24 cycles. Vaccine administration site was the proximal thigh.
  Other Names: CAP1-6D
  Arms: C: CEA peptide 1000mcg

SUMMARY:
The purpose of this study is to determine whether the experimental vaccine "modified CEA peptide CAP 1 -6D" (mCEA) can produce an immune response in patients with pancreatic cancer who have received chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
PC has a dismal prognosis. Despite surgery, chemotherapy, and radiation, most patients with PC will die of distant metastatic disease. Peptide vaccine approaches offer an attractive potential treatment option.

Since CEA is expressed in >90% of PC, it would make an attractive target for a vaccination approach. Several different vaccination approaches have been tested using CEA as a TAA. Although some investigators suggest that DC-based approaches are the most active, they are limited by the need to obtain patient-specific DCs. One attractive approach would be to add GM-CSF to the peptide to recruit endogenous DC to the site of vaccination.

There are data on the use of tumor vaccines in advanced PC. Gjerertsen et al. used a K Ras peptide and GM-CSF in 48 patients with advanced PC. 50% of patients showed a peptide specific CTL response (Gjertsen, Buanes et al. 2001). Those that had an immune response had an increased overall survival, The data from phase I and II clinical trials was based on heavily pretreated patients with metastatic disease. The majority of clinical responses have been disease stabilization. The data in B cell lymphoma vaccines suggests that immune responses are more likely to be generated in minimum disease states (Bendandi, Gocke et al. 1999).

For patients that have had a complete resection and treatment with adjuvant chemoradiation, and for patients with locally advanced nonresectable disease treated with standard chemoradiation, there is presently no therapy available to decrease the chance of disease reoccurrence. Our hypothesis is that immunization with a modified CEA peptide in Montanide/GM-CSF can lead to expansion of CEA-reactive CTL and result in control of CEA expressing pancreatic carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients must express HLA-A2
* Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas that expresses CEA either by IHC or serology.
* Patients prior chemotherapy must have been completed at least 28 days prior to the start of treatment Patients must have completely resected disease or unresectable locally advanced disease.
* Patients with resected disease who had a pancreaticoduodenectomy with negative margins.
* Patients with locally advanced disease or metastatic disease
* Patients must have completed 5FU based chemoradiation>4 weeks, but no more than 12 weeks prior to study registration.
* Age >18 years.
* ECOG performance status 0-1
* Life expectancy greater than 3 months
* Patients must have normal organ and marrow function
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy, biologic therapy, radiotherapy, or an experimental (investigational) agent within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting treatment or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not have received a previous CEA vaccine.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CEA, Montanide ISA-51, or GM-CSF.
* Patients must not have known autoimmune disorders (SLE, Rheumatoid Arthritis), conditions of immunosuppression (such as HIV), or treatment with immunosuppressive drugs (including oral steroids, continuous use of topical steroids, steroid inhalers). Replacement doses of steroids for patients with adrenal insufficiency are allowed.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active GI bleeding, inflammatory bowel disease or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast-feeding women are excluded from this study because peptide vaccines and/or GM-CSF have an unknown effect on a fetus. Breastfeeding should be discontinued if the mother is gong to be treated on this clinical trial.
* Because the risk to patients with immune deficiency treated with peptide vaccine is unknown, HIV-positive patients are excluded from the study. Appropriate studies will be undertaken in patients with intrinsic immunosuppression when indicated.
* Patients with a currently active second malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix are not to be registered. Patients are not considered to have a "currently active" malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-04; Primary Completion 2009-06 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Geynisman DM, Zha Y, Kunnavakkam R, Aklilu M, Catenacci DV, Polite BN, Rosenbaum C, Namakydoust A, Karrison T, Gajewski TF, Kindler HL. A randomized pilot phase I study of modified carcinoembryonic antigen (CEA) peptide (CAP1-6D)/montanide/GM-CSF-vaccine in patients with pancreatic adenocarcinoma. J Immunother Cancer. 2013 Jun 27;1:8. doi: 10.1186/2051-1426-1-8. eCollection 2013. PMID 24829746

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 66 patients screened between August 2004 and September 2009
Period: Overall Study
Arm/Group | A: CEA Peptide 10mcg | B: CEA Peptide 100 mcg | C: CEA Peptide 1000mcg
Started | 7 | 10 | 6
Received at Least 3 Doses of CEA Vaccine | 5 (This group of patients were evaluable for the primary outcome.) | 5 (This group of patients were evaluable for the primary outcome.) | 4 (This group of patients were evaluable for the primary outcome.)
Completed | 5 (2 patients not completing study were randomized but never treated) | 8 (2 patients not completing study were randomized but never treated) | 6
Not Completed | 2 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The 19 patients who received at least 1 dose of the CEA vaccine are included in the baseline analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | A: CEA Peptide 10mcg | B: CEA Peptide 100 mcg | C: CEA Peptide 1000mcg | Total
Number analyzed (Participants) | 5 | 8 | 6 | 19
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 71] | 57.5 [50 to 86] | 61.5 [47 to 77] | 60 [27 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 1 | 4 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 6 | 19
Performance Status [Number; unit: participants] — ECOG performance status scores on a scale from 0-5, with 0 denoting Asymptomatic (Fully active, able to carry on all predisease activities without restriction) and 5 death
  participants
    0 | 2 | 4 | 4 | 10
    1 | 3 | 4 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum T Cell Response From Baseline
Description: T cell frequency (spots per 10^4 CD8+ cells) was measured by ELISPOT (Enzyme-linked immunosorbent spot) assay. Blood was collected for this assay at baseline and every 4 weeks for the first 8 cycles. After the eighth cycle, a blood sample was collected at the time of disease progression. The maximum T cell response was calculated as: peak value on treatment - baseline value.
  A positive value indicates an increase from baseline.
Time Frame: baseline and every 4 weeks on treatment
Population: The analysis population for the primary outcome included the 14 patients who received at least 3 doses of the CEA vaccine and had a ELISPOT at least at baseline and after the 3rd cycle.
Measure: Median (Full Range); unit: spots per 10^4 CD8+ cells
Arm/Group | A: CEA Peptide 10mcg | B: CEA Peptide 100 mcg | C: CEA Peptide 1000mcg
Number analyzed (Participants) | 5 | 5 | 4
spots per 10^4 CD8+ cells | 10.5 [0 to 155] | 51.75 [-16 to 432.5] | 270.625 [72.25 to 377.25]
Statistical Analysis 1: Comparison: A: CEA Peptide 10mcg vs C: CEA Peptide 1000mcg; Test type: Superiority or Other; p = 0.028, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Evidence of Dose Limiting Toxicities of Immunization With Modified CEA (Carcinoembryonic Antigen) Peptide.
Description: Dose-limited toxicity included Grade 2 or higher hemorrhage or allergic reaction or clinical evidence of autoimmune disease. Toxicities were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v2.0.
Time Frame: participants were followed while they were on study treatment, a median of 8 weeks
Measure: Number; unit: participants
Arm/Group | A: CEA Peptide 10mcg | B: CEA Peptide 100 mcg | C: CEA Peptide 1000mcg
Number analyzed (Participants) | 5 | 8 | 6
participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: A: CEA Peptide 10mcg vs B: CEA Peptide 100 mcg vs C: CEA Peptide 1000mcg; Test type: Superiority or Other; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: during study treatment, a median of 8 weeks
Description: Adverse events of grade 2 or higher are reported
Arm/Group | A: CEA Peptide 10mcg | B: CEA Peptide 100 mcg | C: CEA Peptide 1000mcg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 3/5 | 2/8 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: CEA Peptide 10mcg (N=5) | B: CEA Peptide 100 mcg (N=8) | C: CEA Peptide 1000mcg (N=6)
Nausea/vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1
Pain (General disorders) | 2 | 2 | 1
Fatigue (General disorders) | 2 | 2 | 1
Induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes